CLINICAL TRIAL: NCT02337335
Title: Assesment of a Predictive Model Dosage of EPO in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NephroCare Spain (Industry)
Collaborators: Francesc Moreso (Unknown)
Responsible Party: Principal Investigator, Rosa Ramos, Medical Department Management, NephroCare Spain
Other Study IDs: NCSRR01
Record Dates: First submitted 2014-11-03; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Anemia
Keywords: Hemodialyisis; Predictive Model; ESAs; patients
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Assesment of a predictive model of anemia management: Dosage of erythropoietin (EPO) and Iron adminsitration in hemodialysis patients.

DETAILED DESCRIPTION:
Anemia in patients on hemodialysis (HD ) is common and although usually responds well to treatment with Erythropoiesis Stimulating Agents (ESAs ) , this dosage , based on different clinical protocols , often ignores the high variability inter- and intra -individual in patient response . The result leads to swings in the objective by different dosage range that is associated with multiple risks and side effects. There are artificial intelligence-based optimization methods that predict treatment with ESAs in maintaining patient hemoglobin target range . So far the model has been validated for the long half-life of EPO ( darbepoetin ) with promising results.

HYPOTHESIS: Maintaining patients in Hb levels ESAs range using short half-life , avoid the one hand , the need for transfusions and, secondly , the levels exceeding the upper range ( overshooting ), preventing the onset of a increased cardiovascular risk events.

RELEVANCE:The results allow us to validate the model with short half-life ESAs optimizing the management of anemia and improving comorbidity associated with overdosage.

SUMMARY:

Prospective observational study of paired data. Data obtained from the data base Euclid . Data will be collected by clinical teams according to standard clinical practice. Informed at the time of admission to the clinic consent will be obtained . All patient data including to november 15th 2014 and who have completed the study period to 30 april 2015. The results will be compared with those prior to the patient's inclusion in the study were processed.

To detect a difference of 10% in the percentage of patients in the hemoglobin target range after intervention (from 70% to 80%) we will need a minimum sample size of 268 patients assuming an alpha error of 0.05, a beta error of 0.2 and a correlation between both observations of 0.1.

ELIGIBILITY:
Inclusion Criteria:

* > 18 Years
* > 3 Months on HD / OLHDF
* Treated with ESAs( epoBeta ) from> 3 Months

Exclusion Criteria:

* Chronic inflammatory diseases
* Liver Cirrhosis
* Active Neoplasms
* Immunosuppression or other antiinflammatory medication
* Patients who do not require treatment with ESAs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 268 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Erythropoietin stimulating agents dosage | at six months
  u/kg/week
Intravenous Iron dosage | at six months
  mg/mont

SECONDARY OUTCOMES:
anemia parameters | at six months
  ferritin (µg/l), ESA resistance index, transferrin index (%)
Cardiovascular events | at six months
  hospitalisation (days of hospitalisation), death and death cause,

CONTACTS AND LOCATIONS:
Locations (1):
- NephroCare Spain, Tres Cantos, Madrid, Spain